CLINICAL TRIAL: NCT00005496
Title: Inflammation, Infection, and Future Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5014; R01HL058755 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Cerebrovascular Accident; Myocardial Infarction; Venous Thromboembolism; Heart Diseases; Infection; Chlamydia Infections; Cytomegalovirus Infections; Helicobacter Infections; Herpesviridae Infections; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Stroke; Myocardial Infarction; Venous Thromboembolism; Heart Diseases; Infections; Chlamydia Infections; Cytomegalovirus Infections; Helicobacter Infections; Herpesviridae Infections; Inflammation

SUMMARY:
To examine markers of underlying chronic inflammation and infection as potential risk factors for future myocardial infarction (MI), stroke (CVA), and venous thromboembolism (VTE) in plasma samples collected at baseline from healthy participants in the Physicians' Health Study (PHS).

DETAILED DESCRIPTION:
BACKGROUND:

The PHS is a cohort which included 14,916 men initially free of cardiovascular disease and cancer who provided plasma samples at study entry in 1982. These men were randomly assigned in a factorial design to aspirin or beta-carotene therapy, and have been followed prospectively for the occurrence of vascular disease.

DESIGN NARRATIVE:

Employing a nested case-control design, baseline plasma samples are assayed for four markers of inflammation (interleukin-6, TNF-alpha, soluble ICAM, soluble VCAM) and four markers of chronic infection (antibody titers directed against Chlamydia pneumoniae, Helicobacter pylori, Herpes simplex virus, and cytomegalovirus). Case subjects are those study participants who have subsequently developed MI (N=550), CVA (N=400), or VTE (N=200). Control subjects are selected from those study participants who remained healthy during follow-up and are matched to the cases by age, smoking status, and follow-up time. Data on usual cardiovascular risk factors, lipid parameters, and hemostatic markers of risk are already available in the PHS and will be used to evaluate the results for potential confounding and effect modification. Since the PHS was a randomized trial of low-dose aspirin for its initial 5 years, this cohort also provides the unique opportunity to investigate whether the use of an agent with anti-inflammatory properties modifies the risk of subsequent thrombosis among those with underlying inflammation. Indeed, this intriguing hypothesis has recently been raised regarding data relating another marker of inflammation, C-reactive protein, to future risks of myocardial infarction and stroke.

These analyses will take advantage of an existing blood bank from a well-characterized large cohort with many years of follow-up and high quality end-point verification. Thus, this study could provide an efficient and cost-effective mechanism to evaluate the posited, but unproven roles of inflammation and infection as risk factors for future cardiovascular disease.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ridker — Brigham and Women's Hospital

REFERENCES:
- [Background] Ridker PM, Rifai N, Stampfer MJ, Hennekens CH. Plasma concentration of interleukin-6 and the risk of future myocardial infarction among apparently healthy men. Circulation. 2000 Apr 18;101(15):1767-72. doi: 10.1161/01.cir.101.15.1767. PMID 10769275
- [Background] Rifai N, Tracy RP, Ridker PM. Clinical efficacy of an automated high-sensitivity C-reactive protein assay. Clin Chem. 1999 Dec;45(12):2136-41. PMID 10585345
- [Background] Ridker PM, Hennekens CH, Stampfer MJ, Wang F. Prospective study of herpes simplex virus, cytomegalovirus, and the risk of future myocardial infarction and stroke. Circulation. 1998 Dec 22-29;98(25):2796-9. doi: 10.1161/01.cir.98.25.2796. PMID 9860778
- [Background] Blake GJ, Ridker PM. High sensitivity C-reactive protein for predicting cardiovascular disease: an inflammatory hypothesis. Eur Heart J. 2001 Mar;22(5):349-52. doi: 10.1053/euhj.2000.2280. No abstract available. PMID 11207073
- [Background] Zee RY, Bates D, Ridker PM. A prospective evaluation of the CD14 and CD18 gene polymorphisms and risk of stroke. Stroke. 2002 Apr;33(4):892-5. doi: 10.1161/01.str.0000014564.75483.ec. PMID 11935032
- [Background] Liu S, Manson JE, Buring JE, Stampfer MJ, Willett WC, Ridker PM. Relation between a diet with a high glycemic load and plasma concentrations of high-sensitivity C-reactive protein in middle-aged women. Am J Clin Nutr. 2002 Mar;75(3):492-8. doi: 10.1093/ajcn/75.3.492. PMID 11864854
- [Background] Zee RY, Lunze K, Lindpaintner K, Ridker PM. A prospective evaluation of the interleukin-1 receptor antagonist intron 2 gene polymorphism and the risk of myocardial infarction. Thromb Haemost. 2001 Nov;86(5):1141-3. PMID 11816697
- [Background] Albert MA, Rifai N, Ridker PM. Plasma levels of cystatin-C and mannose binding protein are not associated with risk of developing systemic atherosclerosis. Vasc Med. 2001;6(3):145-9. doi: 10.1177/1358836x0100600304. PMID 11789968
- [Background] Blake GJ, Schmitz C, Lindpaintner K, Ridker PM. Mutation in the promoter region of the beta-fibrinogen gene and the risk of future myocardial infarction, stroke and venous thrombosis. Eur Heart J. 2001 Dec;22(24):2262-6. doi: 10.1053/euhj.2001.2692. PMID 11728146
- [Background] Blake GJ, Dada N, Fox JC, Manson JE, Ridker PM. A prospective evaluation of lipoprotein-associated phospholipase A(2) levels and the risk of future cardiovascular events in women. J Am Coll Cardiol. 2001 Nov 1;38(5):1302-6. doi: 10.1016/s0735-1097(01)01554-6. PMID 11691499
- [Background] Chae CU, Lee RT, Rifai N, Ridker PM. Blood pressure and inflammation in apparently healthy men. Hypertension. 2001 Sep;38(3):399-403. doi: 10.1161/01.hyp.38.3.399. PMID 11566912
- [Background] Ridker PM, Danesh J, Youngman L, Collins R, Stampfer MJ, Peto R, Hennekens CH. A prospective study of Helicobacter pylori seropositivity and the risk for future myocardial infarction among socioeconomically similar U.S. men. Ann Intern Med. 2001 Aug 7;135(3):184-8. doi: 10.7326/0003-4819-135-3-200108070-00010. PMID 11487485
- [Background] Pradhan AD, Manson JE, Rifai N, Buring JE, Ridker PM. C-reactive protein, interleukin 6, and risk of developing type 2 diabetes mellitus. JAMA. 2001 Jul 18;286(3):327-34. doi: 10.1001/jama.286.3.327. PMID 11466099
- [Background] Ridker PM, Rifai N, Clearfield M, Downs JR, Weis SE, Miles JS, Gotto AM Jr; Air Force/Texas Coronary Atherosclerosis Prevention Study Investigators. Measurement of C-reactive protein for the targeting of statin therapy in the primary prevention of acute coronary events. N Engl J Med. 2001 Jun 28;344(26):1959-65. doi: 10.1056/NEJM200106283442601. PMID 11430324
- [Background] Zee RY, Lindpaintner K, Struk B, Hennekens CH, Ridker PM. A prospective evaluation of the CD14 C(-260)T gene polymorphism and the risk of myocardial infarction. Atherosclerosis. 2001 Feb 15;154(3):699-702. doi: 10.1016/s0021-9150(00)00698-5. PMID 11257272
- [Background] Redberg RF, Rifai N, Gee L, Ridker PM. Lack of association of C-reactive protein and coronary calcium by electron beam computed tomography in postmenopausal women: implications for coronary artery disease screening. J Am Coll Cardiol. 2000 Jul;36(1):39-43. doi: 10.1016/s0735-1097(00)00680-x. PMID 10898410
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Ridker PM, Hennekens CH, Buring JE, Kundsin R, Shih J. Baseline IgG antibody titers to Chlamydia pneumoniae, Helicobacter pylori, herpes simplex virus, and cytomegalovirus and the risk for cardiovascular disease in women. Ann Intern Med. 1999 Oct 19;131(8):573-7. doi: 10.7326/0003-4819-131-8-199910190-00004. PMID 10523217
- [Background] Ridker PM, Hennekens CH, Rifai N, Buring JE, Manson JE. Hormone replacement therapy and increased plasma concentration of C-reactive protein. Circulation. 1999 Aug 17;100(7):713-6. doi: 10.1161/01.cir.100.7.713. PMID 10449692
- [Background] Blake GJ, Otvos JD, Rifai N, Ridker PM. Low-density lipoprotein particle concentration and size as determined by nuclear magnetic resonance spectroscopy as predictors of cardiovascular disease in women. Circulation. 2002 Oct 8;106(15):1930-7. doi: 10.1161/01.cir.0000033222.75187.b9. PMID 12370215
- [Background] Pradhan AD, Rifai N, Ridker PM. Soluble intercellular adhesion molecule-1, soluble vascular adhesion molecule-1, and the development of symptomatic peripheral arterial disease in men. Circulation. 2002 Aug 13;106(7):820-5. doi: 10.1161/01.cir.0000025636.03561.ee. PMID 12176954
- [Background] Zee RY, Bates D, Ridker PM. A prospective evaluation of the heat shock protein 70 gene polymorphisms and the risk of stroke. Thromb Haemost. 2002 Apr;87(4):622-5. PMID 12008944
- [Background] Zee RY, Ridker PM. Polymorphism in the human C-reactive protein (CRP) gene, plasma concentrations of CRP, and the risk of future arterial thrombosis. Atherosclerosis. 2002 May;162(1):217-9. doi: 10.1016/s0021-9150(01)00703-1. PMID 11947917
- [Background] Zee RY, Hegener HH, Cook NR, Ridker PM. C-reactive protein gene polymorphisms and the risk of venous thromboembolism: a haplotype-based analysis. J Thromb Haemost. 2004 Aug;2(8):1240-3. doi: 10.1111/j.1538-7836.2004.00773.x. PMID 15304023